CLINICAL TRIAL: NCT01884181
Title: Accelerated Diffusion MRI as a Potential Image Based Biomarker for Hungtington Disease
Brief Title: Accelerated Diffusion MRI for Diagnosis of Hungtington Disease
Status: Completed | Type: Observational
Sponsor: Wang . Jiun-Jie (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor-Investigator, Wang . Jiun-Jie, Professor, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Other Study IDs: 102-1056B
Record Dates: First submitted 2013-06-19; First posted 2013-06-21 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Huntington Disease
Keywords: Huntington Disease, diffusion MRI, diagnosis, fast imaging
MeSH Terms: conditions — Huntington Disease; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Huntington Disease Group: Established diagnosis by a neurological examination and genetic assessment of CAG expansion in the Htt gene.
- Healthy Controls: 1. The healthy control subjects without a clinically significant neuropsychiatric disorders.
  2. Able to understand and provide signed informed consent.
  3. Age range and gender matched with Patients with Huntington Disease Group.

SUMMARY:
The hypotheses of the project are

1. Diffusion MRI using compressed sensing could have reduced motion sensitivity and improved susceptibility related artifact because of accelerated acquisition.
2. The macromolecule deposition in the brain of patients with Huntington Disease (HD) can lead to changes detectible by diffusion MRI.

To validate the hypothesis that the new accelerated diffusion MRI technique could produce a new biomarker for HD, patients with Huntington Disease will be recruited. The diffusion index will be calculated using accelerated acquisition. The diagnostic performance will be evaluated for data reconstructed with and without acceleration. The correlation with the disease severity will be assessed.

DETAILED DESCRIPTION:
Diffusion magnetic resonance imaging has emerged as a sensitive, noninvasive tool for assessing the abnormalities in the central nervous system. Applications have been reported in many neurological disorders. However, because of the motion-sensitizing diffusion gradient and the prolonged diffusion encoding time, clinical practice could be difficult especially in patients with motor disorders such as Huntington Disease. Currently there existed no useful biomarker which could reflect either the disease progression or severity of Huntington disease. There is a growing interest in imaging Huntington disease using diffusion magnetic resonance imaging because of its capability to depict the micro-environmental changes.

Unfortunately the excessive motor abnormality such as chorea yields the acquisition of diffusion magnetic resonance imaging unfeasible in a clinical setting. The diffusion MRI with compressed sensing demonstrated reduced motion sensitivity and improved susceptibility related artifact because of the accelerated acquisition. Because of the reduced acquisition time, diffusion MRI in patient with Huntington Disease would be possible. It is therefore expected that the macromolecule deposition in the brain of patients with HD can lead to detectible changes in diffusion properties. The accelerated diffusion MRI techniques will be used to acquire data from healthy volunteers and patients with Huntington disease. The aim of the study is to develop and optimize a novel accelerated diffusion Magnetic Resonance Imaging (MRI) technique using advanced compressed sensing techniques. The joint sparsity constraint algorithm will be implemented in an in-line reconstruction platform for the diffusion MRI processing.

The second aim is to test the efficiency of the new accelerated diffusion MRI technique from phantom and in healthy human. Finally to validate the hypothesis that the new accelerated diffusion MRI technique could produce a new biomarker for HD, patients with Huntington Disease will be recruited. The diffusion index will be calculated using accelerated acquisition. The diagnostic performance will be evaluated for data reconstructed with and without acceleration. The correlation with the disease severity will be assessed. A risk management report will be concluded at the end of project execution for registration in the department of health. The acceleration diffusion MRI could provide new insight to the etiology of the disease. The in-line image reconstruction platform could be used for pediatric or psychiatric patients who cannot hold still in the scanner for a prolonged period and in patients with movement disorders.

ELIGIBILITY:
Inclusion Criteria:

* Huntington Disease

  1. All participants should be aged between 20 and 70 year old.
  2. Established diagnosis by a neurological examination and genetic assessment of CAG expansion in the Htt gene.
  3. Able to understand and provide signed informed consent.
* Healthy Controls:

  1. Able to understand and provide signed informed consent
  2. age range and gender matched with Patients with HD
  3. without significant neuropsychiatric disorders

Exclusion Criteria:

Human Subjects The participants will be divided into 2 groups: Huntington Disease Group and Healthy Control Group. All participants should be aged between 20 and 70 year old, right handed and gender balanced.

Exclusion CriteriaThe following exclusion criteria apply to both groups.

1. Cardiac pacemaker implantation.
2. Implantation of intracranial metal device.
3. Significant major systemic disease, such as renal failure, heart failure, stroke, AMI/unstable angina, poor controlled diabetes mellitus, poor controlled hypertension.
4. Pregnant or breast feeding women.
5. Severe dementia.
6. Any documented abnormality of brain caused by etiologies other than HD by MRI and 18FDG PET studies, which might contribute to the cognitive function, such as hydrocephalus or encephalomalacia, will be excluded. Mild cortical atrophy will be allowed.
7. History of intracranial operation, including thalamotomy, pallidotomy, and/or deep brain stimulation.
8. Significant physical disorder or neuropsychiatric disorder.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Healthy Controls:
     The healthy controls will be recruited from the local community, or the neurological clinic. The cognitive performance will be evaluated by Mini-Mental State Examination (MMSE). A complete physical and neurological examination will be performed.
  2. Huntington Disease:
  Patients with Huntington Disease will be referred from the department of neurology in ChangGung Memorial Hospital, LinKou. Established diagnosis will be made by a neurological examination and genetic assessment of CAG expansion in the Htt gene. The severity and progression of the disease will be assessed by the Unified Huntington's Disease Rating Scale (UHDRS) (18). The cognitive performance will be evaluated by Mini-Mental State Examination (MMSE). The inclusion criteria are the following:
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Feasibility study on healthy human. | the 30th month
  Procedure:
  Diffusion MRI will be acquired form healthy volunteers.
  Approach:
  Images will be acquired with and without compressed sensing DTI The reproducibility of compressed sensing diffusion MRI will be assessed in human

SECONDARY OUTCOMES:
Diagnosis Huntington Disease | end of the fourth year
  Procedure:
  1. Diffusion MRI will be acquired from patients with HD
  2. Diagnostic performance will be analyzed when compared to the healthy control in Validation II in a case control study.
  3. The correlation with disease severity and the image finding will be examined. Approach
  1. ROI selected from basal ganglia 2. The receiver operative characteristic analysis will be performed and the area under curve will be determined. 3. The disease severity will be assessed by Unified Huntington Disease Scale. The correlation will be assessed by Spearmann's Ranked correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Jiun-Jie Wang, PhD, Principal Investigator — ChangGung University
Locations (1):
- ChangGung Memorial Hospital, Linkou, Taoyuan District, Taiwan